CLINICAL TRIAL: NCT04092140
Title: Neuromuscular Ultrasound Changes in Neuropathies in Correlation to Neurophysiological Findings
Brief Title: Neuromuscular Ultrasound in Correlation to Neurophysiological Findings
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shahera Sayed Ahmed Abd El Maged, Resident doctor at neuropsychiatry department, Assiut University
Other Study IDs: ultrasound in neuropathies
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Carpal Tunnel Syndrome; Diabetic Neuropathies; Guillain-Barre Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome; Diabetic Neuropathies; Guillain-Barre Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic complaining of neuropathy or not: using of ultrasound in examination and nerve conduction study
  Interventions: Device: ultrasound
- carpal tunnel syndrome: using of ultrasound in examination and nerve conduction study
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — easy new non invasive tool
  Other Names: ultrasonography

SUMMARY:
1. Study the neuromuscular ultrasound findings in different types of neuropathies
2. correlation between ultrasound and neurophysiological findings in peripheral nerve diseases
3. correlation between clinical pain scale and severity of neuropathy

DETAILED DESCRIPTION:
Ultrasonography is a diagnostic tool that is increasingly used in the work-up of peripheral nerve disease.

As many peripheral nerves run a superficial course, especially in the arms. This is a big advantage over Magnetic Resonance Imaging that is relatively expensive, time consuming and not readily available everywhere.

Nerve cross-sectional area (CSA) can be determined at multiple sites along the nerve.

CSA can be measured at entrapment sites but also at nonentrapment sites. vascularization, echogenicity, fascicular pattern and endoneurial thickness can be investigated as well. All those modalities can give critical insight in the origin and development of various peripheral neuropathies1,2,3

Major peripheral nerves in the extremities, such as the median,ulnar thick enough to reflect the sound beam, resulting in hyperechoic on the US scan 4.

The correlation between nerve conduction study parameters and CSA in ultrasound Ultrasound of the peripheral nervous system is an additional useful diagnostic tool in neuromuscular disorders..5,6,7,8,9 In the longitudinal plane, nerves present as long, slim structures with a mixture of parallel hypoechoic and hyperechoic lines.

Nerves must be distinguished from other nearby structures to ensure correct identification Muscles are hypoechoic and interspersed with small hyperechoic foci which easily distinguishes muscles from nerves. Tendons, which are sometimes adjacent to nerves, move proportionately with joint movement.

US has higher specificity than sensitivity in differentiating myopathic and neuropathic changes The most sensitive diagnostic marker for symptomatic carpal tunnel syndrome patients is an enlarged crosssectional area of the median nerve 10,11,12

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old
* males or females
* diabetic complaining of neuropathy or not
* carpal tunnel syndrome
* Guillain-Barré syndrome

Exclusion Criteria:

* Patient refuse to participate
* The anatomy is altered due to sever trauma,tumor,or surgery
* Severe spasticity preventing examination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Setting:in assuit university hospitals, neuropsychiatry hospital,neurology, orthopedic ,and internal medicine outpatients clinics subjects:will include two groups : peripheral nerve diseases group and healthy control group
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Nerve ultrasound | 3 years
  on median and ulnar nerves
muscle Ultrasound | 3 years
  on thenar and hypothenar muscles
nerve conduction studies | 3 years
  for median and ulnar nerves (sensory and motor)
Electromyogram | 3 years
  for thenar and hypothenar